CLINICAL TRIAL: NCT01364077
Title: Efficacy and Safety of Ivabradine in Hemodialysed Patients With Increased Heart Rate
Brief Title: Ivabradine in Hemodialysed Patients With Increased Heart Rate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Gennaro Cice, MD, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IV-DIAL.01; IV-DIAL.01-A (Other: Second Univesity of Naples)
Record Dates: First submitted 2011-05-25; First posted 2011-06-02 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: High Heart Rate
Keywords: Heart rate; Dialysis; ESRD; ivabradine
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivabradine (Active Comparator)
  Interventions: Drug: Ivabradine
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine — Ivabradine 5 mg BID titrated to 7.5 mg if tolerated
  Arms: Ivabradine
Drug: Placebo — Matched placebo
  Arms: Control

SUMMARY:
A significant association between resting heart rate (HR) and both all-cause mortality and cardiovascular mortality has been demonstrated in numerous epidemiologic studies for both the general population and for patients with cardiovascular disease.

Cardiac disease is the leading cause of death among hemodialysis (HD) patients a recent study reported that the 48-hr mean HR is an independent predictor of cardiovascular events in normotensive hemodialysis patients.

Ivabradine, a pure HR lowering agent,acting on If current inhibition has proven beneficial antianginal effects and mortality reduction linked to HR reduction in ischemic patients.

Aim:

To evaluate the safety and efficacy of ivabradine in normotensive hemodialysed patients with increased pre-dialysis HR (> 80 bpm)

ELIGIBILITY:
Inclusion Criteria:

* Dialysis patients
* Sinus rhythm
* Pre-dialytic Heart rate > 80 bpm

Exclusion Criteria:

* Atrial fibrillation/atrial flutter
* Heart failure
* Valvular disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Heart rate | 1 year

SECONDARY OUTCOMES:
Number of patients that experienced hypotension | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Cice, MD, Principal Investigator — Second Univesity of Naples
Locations (1):
- Chair of Cardiology, Naples, Italy